CLINICAL TRIAL: NCT05193916
Title: A Multi-Center, Randomised, Double-blind, Placebo Controlled Phase II Clinical Study of Chiglitazar in Patients With Nonalcoholic Steatohepatitis Accompanied by Elevated Triglycerides and Insulin Resistance
Brief Title: A Phase II Clinical Trial of Chiglitazar for NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CGZ203; CINAR (Other: Chipscreen)
Record Dates: First submitted 2021-12-03; First posted 2022-01-18 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: NASH

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chiglitazar low dose (Experimental): 3 tablets of drug and 1 tablet of placebo p.o. per day
  Interventions: Drug: chiglitazar sodium tablets
- Chiglitazar high dose (Experimental): 4 tablets p.o. per day
  Interventions: Drug: chiglitazar sodium tablets
- control group (Placebo Comparator): 4 placebo tablets p.o. per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: chiglitazar sodium tablets — the drugs will be given orally once a day
  Other Names: Bilessglu®; CS-038; Carfloglitazar
  Arms: Chiglitazar high dose; Chiglitazar low dose
Drug: Placebo — no active drug contained
  Other Names: simulant of chiglitazar
  Arms: control group

SUMMARY:
The study is to evaluate the efficacy and safety of chiglitazar monotherapy in patients with non-clcoholic steatohepatitis (NASH).

DETAILED DESCRIPTION:
The study is a non-invasive exploratory phase II trial in patients who were clinically diagnosed as non-alcoholic steatohepatitis (NASH) with liver fibrosis accompanied by elevated triglycerides (TG) and insulin resistance. The efficacy and safety of chiglitazar tablets 48mg and 64mg will be compared with placebo in the 18-week-treament.

ELIGIBILITY:
Inclusion Criteria:

1. Before any evaluation, an informed consent form voluntarily signed by the patient must be obtained;
2. 18 -75 years old (at the time of screening visit V1), male or female;
3. MRI-PDFF ≥ 8% ;
4. Liver stiffness value ( LSM ) 7.0-11.0kPa ;
5. Triglyceride ( TG ) ≥1.7mmol/L and ≤5.6 mmol/L;
6. HOMA-IR ≥ 2.5 ;
7. Serum Alanine aminotransferease (ALT) ≥ the upper limit of normal during screening.

Exclusion Criteria:

1. Type 1 diabetes;
2. Any of the following for type 2 diabetes:

   * HbA1c ≥ 8.5% during screening
   * At the time of screening, ≥ 2 oral hypoglycemic drugs combinations
   * Receiving any of the following medications at screening: Thiazolidinediones (TZD) drugs, fibrates, glucagon-like peptide-1 (GLP-1) receptor agonists, insulin
3. Existing other liver diseases or history of liver diseases
4. History of transient ischemic attack or cerebrovascular accident;
5. History of myocardial infarction, or coronary angioplasty or coronary artery bypass surgery, unstable angina, heart failure (New York Heart Association NYHA grade III / IV ), or ECG signs of left ventricular hypertrophy, or serious arrhythmias ；
6. During screening, blood pressure ≥ 160/100 mmHg ;
7. Previous or planned ( during the study period) bariatric surgery;
8. Liver transplantation history or planned liver transplantation;
9. Liver biopsy show liver cirrhosis or clinically diagnosed as cirrhosis;
10. Weight loss of more than 5% in 6 months before screening;
11. History of edema of lower limbs or whole body;
12. diagnosed as osteoporosis or any other known bone disease;
13. Donated blood or lost blood >400 ml within 8 weeks before the first medication;
14. With MRI scan contraindications;
15. In the past 5 years, there was a history of malignant tumors of any organ system;
16. Human immunodeficiency virus ( HIV ) test is positive;
17. Heavy drinking of alcohol for more than 3 months in a year;
18. Heavy smoking >30 per day within 1 year;
19. History of drug abuse in 12 months;
20. Drugs cumulatively for more than 1 month in the previous 3 months before screening, such as obeticholic acid ( OCA ), berberine;
21. Drugs that may cause liver damage for more than 2 weeks within 1 year before screening;
22. Patients received the following medications unless they have received a stable dose for at least 1 month before screening :Beta-blockers, thiazide diuretics, statins, niacin, ezetimibe, thyroid hormone;
23. The calculated eGFR < 60 mL/(min*1.73m^2 );
24. There is clinical evidence of liver decompensation or severe liver damage;
25. Low density lipoprotein cholesterol (LDL-C) ≥ 3.4 mmol/L during screening ;
26. Platelet < 100×10^9 /L ;
27. Patient participating in other clinical trials of drugs or medical devices within 3 months prior to screening ;
28. Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline to week 18 in liver fat content as measured by MRI using the proton density fat fraction (MRI-PDFF) | 18 weeks
  center reading for the primary endpoint

SECONDARY OUTCOMES:
the change in liver fat content from baseline as shown by MRI-PDFF after 18 weeks treatment | 18 weeks
  Absolute decrease in liver fat content Proportion of patients with Liver fat content absolute decrease ≥5% Proportion of patients with Liver fat content relative decrease ≥30% proportion
ALT changes from baseline | 6,12,18 weeks
  changes from baseline in liver enzymes
FIB-4 changes from baseline | 6,12,18 weeks
  changes from baseline in Fibrosis 4 Score
insulin resistance changes | 6,12,18 weeks
  Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)
Changes from baseline in TG | 6,12,18 weeks
  blood sample
change from baseline in Liver stiffness measurement (LSM) with Fibroscan | 6,12,18 weeks
  to evlaute the severity of liver fibrosis
change from baseline in Cytokeratin18 (CK-18) | 6,12,18 weeks
  to evaluate the severity of liver damage
Maximum Plasma Concentration [Cmax] of chiglitazar after 1 dose, 6 weeks and 12 weeks of treatment | 0, 6,12 weeks
  population PK
The area under the plasma drug concentration-time curve [AUC] of chiglitazar after 1 dose, 6 weeks and 12 weeks of treatment | 0, 6,12 weeks
  population PK

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Foshan First People's Hospital, Foshan, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Jiangsu
  - Nanjing Second Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Ch’ang-ch’un, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shanghai Tongren Hospital, Shanghai, Shanghai Municipality
  - The Ninth People's Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No